CLINICAL TRIAL: NCT03917498
Title: Single Pre-Operative Radiation Therapy - With Delayed Surgery (SPORT-DS) for Low Risk Breast Cancer: A Phase 1 Study
Brief Title: Single Pre-Operative Radiation Therapy - With Delayed Surgery for Low Risk Breast Cancer
Acronym: SPORT-DS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Yassa (Other)
Responsible Party: Sponsor-Investigator, Michael Yassa, Radiation Oncologist, Maisonneuve-Rosemont Hospital
Organization: Maisonneuve-Rosemont Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPORT-DS
Record Dates: First submitted 2019-04-11; First posted 2019-04-17 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
Keywords: radiation therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Pre-Operative Radiation Therapy with Delayed Surgery (Experimental): Single Pre-Operative Radiation Therapy with Delayed Surgery
  Interventions: Radiation: Single Pre-Operative Radiation Therapy - with Delayed Surgery

INTERVENTIONS:
Radiation: Single Pre-Operative Radiation Therapy - with Delayed Surgery — Single Pre-Operative Radiation Therapy - with Delayed Surgery

SUMMARY:
To study a single dose of preoperative partial radiotherapy to a low-risk breast tumour. The radiotherapy will be goven 3 months before surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged 65 years or older
2. World Health Organization (WHO) performance status 0-2
3. Invasive ductal carcinoma proven by biopsy done ≤ 12 weeks from treatment start
4. Unifocal disease on preoperative staging ultrasound done ≤ 12 weeks from treatment start
5. Tumors less than 2cm clinically on physical exam, as well as on breast ultrasound
6. No clinical evidence of nodal disease (i.e. cN0), on physical examination done ≤ 12 weeks from treatment start, as well as on breast ultrasound
7. Estrogen receptor status (ER) positive on biopsy
8. Her2 negative on biopsy
9. Grade 1 or 2 on biopsy
10. Planned surgery is a partial mastectomy with sentinel lymph node biopsy
11. Localisation markers placed before treatment

Exclusion Criteria:

1. Age less than 65 years
2. A known deleterious mutation in BRCA 1 and/or BRCA 2
3. Clinical tumor size > 2.0 cm in greatest diameter on staging ultrasound
4. Tumor histology limited to lobular carcinoma only
5. Clinically positive axillary nodes (cN+)
6. Lymphovascular invasion on biopsy
7. Pure ductal or lobular carcinoma in situ on biopsy
8. Extensive intraductal component on biopsy
9. Neoadjuvant hormonal manipulation or chemotherapy
10. Prior history of cancer (Patients with prior or concurrent basal cell or squamous cell skin cancers are eligible for the trial)
11. More than one primary tumor in different quadrants of the same breast
12. Diffuse microcalcifications on mammography
13. Paget's disease of the nipple
14. Previous irradiation to the ipsilateral breast
15. Presence of an ipsilateral breast implant or pacemaker
16. Serious non-malignant disease (e.g. cardiovascular, pulmonary, systemic lupus erythematosus (SLE), scleroderma) which would preclude definitive radiation treatment
17. Estrogen receptor status (ER) not known
18. Currently pregnant or lactating
19. Psychiatric or addictive disorders which would preclude obtaining informed consent or adherence to protocol
20. Geographic inaccessibility for follow-up
21. Lack of preoperative staging with breast and axillary ultrasound
22. Inability to adequately plan the patient for the experimental technique

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
rate of pathological complete response | at the time of surgery

SECONDARY OUTCOMES:
incidence of radiation toxicity | in the 2 years after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Lavigne D, Hijal T, Vavassis P, Guilbert MC, Sideris L, Dube P, Gervais MK, Leblanc G, Dufresne MP, Nguyen D, Tiberi D, Mahmoud D, Yassa M. Single preoperative radiation therapy with delayed surgery for low-risk breast cancer: Oncologic outcome, toxicity and cosmesis of the SPORT-DS phase I trial. Radiother Oncol. 2024 Nov;200:110515. doi: 10.1016/j.radonc.2024.110515. Epub 2024 Aug 30. PMID 39218041